CLINICAL TRIAL: NCT02915029
Title: Reducing Health Disparity in Chronic Kidney Disease in Zuni Indians
Brief Title: Home-base Kidney Care in Zuni Indians
Acronym: HBKC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Zuni Tribal Administration (Unknown); Zuni comprehensive Community Health Center, Indian Health Services (Unknown)
Responsible Party: Principal Investigator, Vallabh O Shah, Professor, University of New Mexico
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-249 -sub study HBKC
Record Dates: First submitted 2016-09-08; First posted 2016-09-26 (Estimated); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-04 (Actual); Status verified 2019-12

CONDITIONS: Chronic Kidney Disease
Keywords: Native American; Community Health Representative; Home base; Diabetes; Point of care testing; Patient Activation Measure; Patient preferences
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Patient Preference

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Education and Lifestyle Coaching (Experimental): Education and life style coaching includes:
  education about diabetes and kidney disease Coaching /counseling about lifestyle, nutrition and medication adherence
  Interventions: Other: Educational and lifestyle coaching
- Usual care (UC) control arm (No Intervention): once randomize to the Usual Care control group, the participants are left alone and are suggested to contact their providers for health care. The group gets labs and other survey done at 6 and 12 months of the intervention.

INTERVENTIONS:
Other: Educational and lifestyle coaching — Educational lifestyle and patient activation is a CHR lead home visits every other week to provide education on healthy lifestyles (diet, exercise, alcohol abuse and smoking) as patient preference; Education provided on management of diabetes, hypertension and hyperlipidemia POC testing for A1C and microalbuminuria conducted at patient homes. Lifestyle and diet related Motivational messaging carried out regularly. Patient will receive group session at the clinic every quarters.
  Control arm will receive their usual care provided by IHS. The control group will receive a health evaluation at the initiation of the study and at the 6-month and 12-month.
  Arms: Education and Lifestyle Coaching

SUMMARY:
People reach End Stage Renal Disease (ESRD) due to progressive chronic kidney disease (CKD). CKD is associated with increased risks for heart disease and death. The burden of chronic kidney disease is increased among minority populations compare to Caucasians. The Zuni Indians are experiencing an epidemic of chronic kidney disease is due primarily to the high rates of obesity and diabetes. The present study entitled Home-Based Kidney Care is designed to delay / reduce rate of ESRD by early interventions in CKD. Investigators propose to assess the safety and efficacy of conducting a full-scale study to determine if home based care delivered by a collaborative team composed of community health workers and University of New Mexico faculty will decrease the risk for the development and the progression of CKD.

DETAILED DESCRIPTION:
Hypothesis: (1) The Zuni Health Initiative (ZHI) can integrate an innovative approach to Home based kidney care (HBKC) utilizing tribal Community Health Representatives (CHRs), Point of Care (POC) technology, telemedicine and motivational messaging in conjunction with patient preferences and Patient Activation Measures (PAM) into the chronic care model to improve the detection and treatment of Chronic Kidney Disease (CKD) and related risk factors; (2) This model is generalizable to other high-risk communities e.g., Hispanic and American Indians in Guadalupe, AZ being studied by NIDDK, NIH-Phoenix.

Specific Aim 1: Re-phenotype prior participants, to identify incident cases of CKD, estimate progression rates, and identify participants for the proposed study of HBKC;

Specific Aim 2: Conduct a pilot study of HBKC in 120 people. Randomize households in a 1:1 allocation to usual care versus HBKC. Compare the changes in Patient Activation measure (PAM), Adherence, BP, weight, HbA1c, UACR, eGFR and lipid profiles between the two groups over the 1-year intervention period;

Specific Aim 3: Inform the design of the full-scale study by estimating anticipated recruitment, adherence and dropout rates, sample size and reassessing the approach;

Specific Aim 4: Assess the exportability of the HBKC model to Hispanics and American Indians in Guadalupe, AZ.

Study Outcomes: (1) The PAM and adherence; (2) Changes in clinical phenotypes including Cr, UACR, A1c, body weight, BMI, fasting glucose, blood pressure (BP), plasma lipids, and inflammatory markers; (3) Changes in the quantitative traits such as diet and scores from a battery of mental-health, self-efficacy, and quality of life instruments.

Health Impact: The active participation of the Zuni tribal leadership and IHS in this protocol, and the general affordability of Zuni native CHR personnel, render the outcomes that will be demonstrated by this proposal easily sustainable over the long term. If successful, this program has the potential to change best-practices for CKD progression and to reduce health disparities in a cost-effective and sustainable manner.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of diabetes
* Clinical diagnosis of microalbuminuria
* Must be living in a household with more than 1 living participant
* Age 21 to 80 years
* Must have negative pregnancy test in women of child-bearing potential

Exclusion Criteria:

* Life expectancy < 1 year
* On dialysis
* With renal transplant
* Pregnancy or absence of reliable birth control in women of child-bearing potential
* Malignancy except non-melanoma skin cancer
* Blind
* Unwilling or unable to give informed consent.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-10; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data will be available to share once the Zuni tribal leadership approves it.

REFERENCES:
- [Background] Shah VO, Carroll C, Mals R, Ghahate D, Bobelu J, Sandy P, Colleran K, Schrader R, Faber T, Burge MR. A Home-Based Educational Intervention Improves Patient Activation Measures and Diabetes Health Indicators among Zuni Indians. PLoS One. 2015 May 8;10(5):e0125820. doi: 10.1371/journal.pone.0125820. eCollection 2015. PMID 25954817
- [Background] Newman S, Cheng T, Ghahate DM, Bobelu J, Sandy P, Faber T, Shah VO. Assessing knowledge and attitudes of diabetes in Zuni Indians using a culture-centered approach. PLoS One. 2014 Jun 11;9(6):e99614. doi: 10.1371/journal.pone.0099614. eCollection 2014. PMID 24919064
- [Background] Shah VO, Ghahate DM, Bobelu J, Sandy P, Newman S, Helitzer DL, Faber T, Zager P. Identifying barriers to healthcare to reduce health disparity in Zuni Indians using focus group conducted by community health workers. Clin Transl Sci. 2014 Feb;7(1):6-11. doi: 10.1111/cts.12127. Epub 2013 Nov 8. PMID 24528897
- [Background] MacCluer JW, Scavini M, Shah VO, Cole SA, Laston SL, Voruganti VS, Paine SS, Eaton AJ, Comuzzie AG, Tentori F, Pathak DR, Bobelu A, Bobelu J, Ghahate D, Waikaniwa M, Zager PG. Heritability of measures of kidney disease among Zuni Indians: the Zuni Kidney Project. Am J Kidney Dis. 2010 Aug;56(2):289-302. doi: 10.1053/j.ajkd.2010.03.012. Epub 2010 Jun 19. PMID 20646805
- [Background] Nelson RG, Pankratz VS, Ghahate DM, Bobelu J, Faber T, Shah VO. Home-Based Kidney Care, Patient Activation, and Risk Factors for CKD Progression in Zuni Indians: A Randomized, Controlled Clinical Trial. Clin J Am Soc Nephrol. 2018 Dec 7;13(12):1801-1809. doi: 10.2215/CJN.06910618. Epub 2018 Nov 15. PMID 30442864
- [Result] Cukor D, Cohen LM, Cope EL, Ghahramani N, Hedayati SS, Hynes DM, Shah VO, Tentori F, Unruh M, Bobelu J, Cohen S, Dember LM, Faber T, Fischer MJ, Gallardo R, Germain MJ, Ghahate D, Grote N, Hartwell L, Heagerty P, Kimmel PL, Kutner N, Lawson S, Marr L, Nelson RG, Porter AC, Sandy P, Struminger BB, Subramanian L, Weisbord S, Young B, Mehrotra R. Patient and Other Stakeholder Engagement in Patient-Centered Outcomes Research Institute Funded Studies of Patients with Kidney Diseases. Clin J Am Soc Nephrol. 2016 Sep 7;11(9):1703-1712. doi: 10.2215/CJN.09780915. Epub 2016 May 19. PMID 27197911

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Number of home visit
Groups:
- Education and Lifestyle Coaching: Education and life style coaching includes:
  education about diabetes and kidney disease Coaching /counseling about lifestyle, nutrition and medication adherence
  Educational and lifestyle coaching: Educational lifestyle and patient activation is a CHR lead home visits every other week to provide education on healthy lifestyles (diet, exercise, alcohol abuse and smoking) as patient preference; Education provided on management of diabetes, hypertension and hyperlipidemia POC testing for A1C and microalbuminuria conducted at patient homes. Lifestyle and diet related Motivational messaging carried out regularly. Patient will receive group session at the clinic every quarters.
  Control arm will receive their usual care provided by IHS. The control group will receive a health evaluation at the initiation of the study and at the 6-month and 12-month.
Period: Overall Study
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Started | 63; 24 Number of home visit | 62; 0 Number of home visit
Completed | 50; 24 Number of home visit | 48; 0 Number of home visit
Not Completed | 13; 0 Number of home visit | 14; 0 Number of home visit

BASELINE CHARACTERISTICS:
Population: Members of the Zuni Pueblo, NM who have evidence of chronic kidney disease based on microalbuminuria of >30 mg/g
Groups:
- Total: Total of all reporting groups
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm | Total
Number analyzed (Participants) | 63 | 62 | 125
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (11) | 48 (12) | 47 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 26 | 57
  Male | 32 | 36 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 63 | 62 | 125
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 63 | 62 | 125
Patient Activation Measure - Total Score [Mean (Standard Deviation); unit: Score] — PAM is 13 questionnaire use a categorical agreement scale with 4 response options: strongly disagree, disagree, agree, strongly agree, and N/A. The raw score is calculated by adding responses to the 13 questions. If all questions are answered, the range of raw scores is from 13 to 52. If there is at least 1 item with a response of N/A, the total score is divided by the number of items completed and multiplied by 13 to yield a normalized raw score.
  The score converts raw scores to an "activation score," ranging from 0 to 100 with a classification level between 1 and 4
  Score | 60.7 (20.5) | 65.1 (14.6) | 62.9 (17.8)
Patient activation level >3 [Number; unit: participants with diabetes] — Number of participants "activated" to be engaged in their own health care.
  participants with diabetes | 43 | 52 | 95
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 129 (17) | 132 (19) | 130 (18)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 83 (13) | 85 (13) | 84 (13)
HbA1c [Mean (Standard Deviation); unit: percentage] — Glycosylated Hemoglobin
  percentage | 7.5 (2.6) | 7.5 (2.3) | 7.5 (2.5)
Hypertension [Count of Participants; unit: Participants] | 36 | 42 | 78
Diabetes status [Count of Participants; unit: Participants] — Count of Participants are with diabetes
  Participants | 33 | 39 | 72
High School Graduate [Count of Participants; unit: Participants] | 41 | 37 | 78
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 32 (8) | 32 (7) | 32 (8)
Serum Total Protein [Mean (Standard Deviation); unit: g/dl] | 7.7 (0.6) | 7.6 (0.6) | 7.7 (0.6)
Serum Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 201 (58) | 181 (38) | 191 (49)
Serum LDL Cholesterol [Mean (Standard Deviation); unit: mg/dl] | 117 (42) | 109 (32) | 113 (37)
Serum HDL Cholesterol [Median (Inter-Quartile Range); unit: mg/dl] | 46 [39 to 62] | 50 [39 to 63] | 48 [39 to 62]
Serum Triglycerides [Median (Inter-Quartile Range); unit: mg/dl] | 139 [100 to 182] | 133 [90 to 200] | 136 [90 to 195]
eGFR [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — Estimated (via CKD-EPI) Glomerular Filtration Rate
  mL/min/1.73 m^2 | 105 (31) | 101 (29) | 103 (30)
UACR [Median (Inter-Quartile Range); unit: mg/g] — Urine Albumin to Creatinine Ratio.
  mg/g | 139 [57 to 377] | 190 [57 to 714] | 155 [57 to 587]
hsCRP [Median (Inter-Quartile Range); unit: mg/L] — High Sensitive c-Reactive Protein
  mg/L | 3.8 [0.9 to 10] | 2.6 [1.3 to 4.1] | 2.9 [1.3 to 6.2]
KDQOL-SP [Mean (Standard Deviation); unit: points] — Symptom/Problem List The KDQOL-36™ is a short form that includes the SF-12 as generic core plus the burden of kidney disease, symptoms/problems of kidney disease, and effects of kidney disease scales from the KDQOL-SF.
  Items 1-12: SF-12 Items 13-16: Burden of kidney disease (k=4) Items 17-28: Symptoms/problems (k=12) Items 29-36: Effects of kidney disease (k=8)
  points | 86.4 (11.2) | 86.6 (14.4) | 86.5 (12.9)
KDQOL-EKD [Mean (Standard Deviation); unit: points] — Effects on Kidney Disease. The KDQOL-36™ is a short form that includes the SF-12 as generic core plus the burden of kidney disease, symptoms/problems of kidney disease, and effects of kidney disease scales from the KDQOL-SF.
  Items 1-12: SF-12 Items 13-16: Burden of kidney disease (k=4) Items 17-28: Symptoms/problems (k=12) Items 29-36: Effects of kidney disease (k=8)
  points | 92.7 (7.3) | 93.2 (12.0) | 92.9 (9.9)
KDQOL-BKD [Mean (Standard Deviation); unit: points] — Burden of Kidney Disease. The KDQOL-36™ is a short form that includes the SF-12 as generic core plus the burden of kidney disease, symptoms/problems of kidney disease, and effects of kidney disease scales from the KDQOL-SF.
  Items 1-12: SF-12 Items 13-16: Burden of kidney disease (k=4) Items 17-28: Symptoms/problems (k=12) Items 29-36: Effects of kidney disease (k=8)
  points | 70.3 (20.5) | 74.3 (23.8) | 72.3 (22.2)
KDQOL-SF12 Physical Score [Mean (Standard Deviation); unit: points] — Physical Score (Quality of Life). The KDQOL-36™ is a short form that includes the SF-12 as generic core plus the burden of kidney disease, symptoms/problems of kidney disease, and effects of kidney disease scales from the KDQOL-SF.
  Items 1-12: SF-12 Items 13-16: Burden of kidney disease (k=4) Items 17-28: Symptoms/problems (k=12) Items 29-36: Effects of kidney disease (k=8)
  points | 45.5 (9.5) | 45.4 (8.5) | 45.5 (9.0)
KDQOL-SF12 Mental [Mean (Standard Deviation); unit: points] — Mental Quality of Life from Short Form-12 The KDQOL-36™ is a short form that includes the SF-12 as generic core plus the burden of kidney disease, symptoms/problems of kidney disease, and effects of kidney disease scales from the KDQOL-SF.
  Items 1-12: SF-12 Items 13-16: Burden of kidney disease (k=4) Items 17-28: Symptoms/problems (k=12) Items 29-36: Effects of kidney disease (k=8)
  points | 47.4 (9.6) | 51.2 (10) | 49.3 (9.8)
Morisky Score [Mean (Standard Deviation); unit: Scores on a scale] — 8-Item Morisky Medication Adherence Scale Morisky Medication Adherence Scale reflect that the reported values are from the 8-item version of the scale: zero remains the lowest level of medication adherence, but 8 is the highest level of medication adherence.
  * The scale of the total score ranges from 0 to 8. We only report a total score.
  * For the reported scale, 0 reflects worse medication adherence and 8 reflects better medication adherence.
  * We didn't combine subscales to compute a total score, but the total score does reflect the number of individual items that were endorsed.
  Scores on a scale | 5.4 (2.3) | 4.6 (2.3) | 5.0 (2.3)

OUTCOME MEASURES:

1. Primary Outcome: Patient Activation Measure (PAM) -13 Item Questionnaire
Description: Patient Activation Measure (PAM) questionnaire gives total score of activation as well as levels (stages) of patient activation.
  PAM total score can range form 0-100 with higher score reflecting higher level of activation in Patient health care.
  PAM levels (Stages) 1 through 4 with 1 being the lowest activation and 4 being the highest activation level.
  We collected data about Changes in PAM score as well as levels (stages) from baseline to 12 months of intervention and compare it to Usual care group.
Time Frame: 12 months follow-up minus baseline values
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 50 | 48
points | 9.1 (26.0) | -1.4 (15.3)
Statistical Analysis 1: Comparison: Education and Lifestyle Coaching; Group 1(usual care) is the comparison group, group 2 is the intervention group; Test type: Superiority — The primary hypothesis being tested was that the intervention will increase patient activation; p = 0.01, ANCOVA; Primary outcome was change in PAM total score, adjusted for baseline level. Adjusting for family clustering with generalized estimated equations; Mean Difference (Net) = 8.7, 95% CI 2-sided [1.9 to 15.5] — This reflects the between-group difference for the within-person change scores in PAM total score adjusting for baseline values per person; Applied generalized estimating equations (GEE) to account for within family (household) clustering

2. Primary Outcome: Patient Activation Measure (PAM) Level Greater Than 2
Description: Participants in an "Activated" category. Patient Activation Measure (PAM) questionnaire gives total score of activation as well as levels (stages) of patient activation.
  PAM total score can range form 0-100 with higher score reflecting higher level of activation in Patient health care.
  PAM levels (Stages) 1 through 4 with 1 being the lowest activation and 4 being the highest activation level. Level 1 labeled as patient being dis-engaged, Level 2 labeled as patient becoming aware of health condition but still struggling, level 3 labeled as patient is taking action and gaining control of their health care and level 4 labeled as maintaining behaviors and pushing forward - for our analysis purposes we classified participants into levels 3 and 4 (activated) and level 1 and 2 as not activated.
  We collected data about Changes in PAM score as well as levels (stages) from baseline to 12 months of intervention and compare it to Usual care group.
Time Frame: 12 months follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 50 | 48
Participants | 44 | 33

3. Secondary Outcome: A1c
Description: Changes in clinical values
Time Frame: 12 months minus baseline values
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 50 | 48
percentage | -0.5 (1.4) | 0.1 (1.4)

4. Secondary Outcome: Diastolic Blood Pressure
Description: Changes in diastolic blood pressure on study.
Time Frame: 12 months minus baseline values
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 50 | 48
mm Hg | -0.1 (12.8) | 0.2 (14.9)

5. Secondary Outcome: Systolic Blood Pressure
Description: Changes in Systolic blood pressure over study.
Time Frame: 12 months minus baseline values
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 50 | 48
mm Hg | 3.4 (19.0) | 5.2 (19.0)

6. Secondary Outcome: Body Mass Index
Description: Changes in the value of body mass index (BMI)
Time Frame: 12 months minus baseline values
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 50 | 48
kg/m^2 | -1.3 (2.1) | -0.2 (1.9)

7. Secondary Outcome: Low-density Lipoprotein LDL Cholesterol
Description: Changes in serum LDL cholesterol on study
Time Frame: 12 months minus baseline values
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 50 | 48
mg/dl | -12.4 (41.2) | -4.9 (36.5)

8. Secondary Outcome: High-density Lipoprotein HDL Cholesterol
Description: Change in serum HDL cholesterol on study
Time Frame: 12 months minus baseline values
Measure: Mean (Inter-Quartile Range); unit: mg/dl
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 50 | 48
mg/dl | 3.5 [-1.8 to 11.8] | 1.5 [-6.0 to 4]

9. Secondary Outcome: Triglycerides
Description: Change in serum triglycerides on study
Time Frame: 12 months minus baseline values
Measure: Median (Inter-Quartile Range); unit: mg/dl
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 50 | 48
mg/dl | -8.0 [-46 to 30.5] | -8.5 [-32.8 to 23.3]

10. Secondary Outcome: Serum Total Cholesterol
Description: Change in total cholesterol on study
Time Frame: 12 months minus baseline values
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 50 | 48
mg/dl | -19 (54.3) | -4.5 (44.5)

11. Secondary Outcome: High Sensitive C-reactive Protein-hsCRP
Description: Changes in the serum c-reactive protein on study
Time Frame: 12 months minus baseline values
Measure: Mean (Inter-Quartile Range); unit: mg/L
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 47 | 46
mg/L | -1.5 [-5.8 to 0] | 1.7 [-0.5 to 6.5]

12. Secondary Outcome: Serum Total Protein
Description: Change in total protein on study
Time Frame: 12 months minus baseline values
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 50 | 47
g/dl | -0.2 (0.4) | -0.1 (0.4)

13. Secondary Outcome: eGFR
Description: Changes in estimated (via CKD-EPI) Glomerular Filtration Rate.
Time Frame: 12 months minus baseline values
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m2
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 50 | 48
mL/min/1.73 m2 | -5.2 (14.2) | -9.6 (12.2)

14. Secondary Outcome: UACR
Description: change in urinary albumin to creatinine ratio on study.
Time Frame: 12 months minus baseline values
Measure: Median (Inter-Quartile Range); unit: mg/g
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 50 | 48
mg/g | -45 [-176 to 13.3] | 17.5 [-62.5 to 359.3]

15. Secondary Outcome: KDQOL-Symptom/Problem
Description: Changes on study of symptom/problem list from quality of life (KDQOL-36). Quality of life (QOL) was measured using the Kidney Disease Quality of Life-36 (KDQOL-36) survey, a kidney-disease-specific quality of life instrument that assesses five domains: general physical health (SF-12 Physical), mental health (SF-12 Mental), burden of kidney disease (BKD), disease symptoms problem list (SP), and effects of kidney disease (EKD). For all KDQOL scales, a higher score indicates better quality of life. All domain scales can range from 0-100.
Time Frame: 12 months minus baseline values
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 47 | 47
points | 0.1 (13.7) | 2.7 (11.5)

16. Secondary Outcome: KDQOL-EKD
Description: Changes in effects of kidney disease score from quality of life (KDQOL). Changes on study of effect of kidney disease from quality of life (KDQOL-36). Quality of life (QOL) was measured using the Kidney Disease Quality of Life-36 (KDQOL-36) survey, a kidney-disease-specific quality of life instrument that assesses five domains: general physical health (SF-12 Physical), mental health (SF-12 Mental), burden of kidney disease (BKD), disease symptoms problem list (SP), and effects of kidney disease (EKD). For all KDQOL scales, a higher score indicates better quality of life. All domain scales can range from 0-100.
Time Frame: 12 months minus baseline values
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 49 | 48
score on a scale | 3.2 (8.0) | 2.9 (8.8)

17. Secondary Outcome: KDQOL-BKD
Description: Change on study of burden of kidney disease score from KDQOL-36. Quality of life (QOL) was measured using the Kidney Disease Quality of Life-36 (KDQOL-36) survey, a kidney-disease-specific quality of life instrument that assesses five domains: general physical health (SF-12 Physical), mental health (SF-12 Mental), burden of kidney disease (BKD), disease symptoms problem list (SP), and effects of kidney disease (EKD). For all KDQOL scales, a higher score indicates better quality of life. All domain scales can range from 0-100.
Time Frame: 12 months minus baseline values
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 49 | 47
score on a scale | 14.8 (22.1) | 2.3 (31.9)

18. Secondary Outcome: KDQOL-SF12 Physical Score
Description: Changes on study of SF12 physical quality of life scale from the KDQOL-36. Quality of life (QOL) was measured using the Kidney Disease Quality of Life-36 (KDQOL-36) survey, a kidney-disease-specific quality of life instrument that assesses five domains: general physical health (SF-12 Physical), mental health (SF-12 Mental), burden of kidney disease (BKD), disease symptoms problem list (SP), and effects of kidney disease (EKD). For all KDQOL scales, a higher score indicates better quality of life. All domain scales can range from 0-100.
Time Frame: 12 months minus baseline values
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 49 | 48
score on a scale | 2.1 (9.4) | 0.8 (10.6)

19. Secondary Outcome: KDQOL-SF12 Mental Score
Description: Change on study of SF12 mental quality of life scale from the KDQOL-36 Quality of life (QOL) was measured using the Kidney Disease Quality of Life-36 (KDQOL-36) survey, a kidney-disease-specific quality of life instrument that assesses five domains: general physical health (SF-12 Physical), mental health (SF-12 Mental), burden of kidney disease (BKD), disease symptoms problem list (SP), and effects of kidney disease (EKD). For all KDQOL scales, a higher score indicates better quality of life. All domain scales can range from 0-100.
Time Frame: 12 months minus baseline values
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 49 | 48
score on a scale | 7.5 (11.0) | -0.2 (10.0)

20. Secondary Outcome: 8-Item Morisky Score
Description: Change in Morisky total score on study.The 8-item Morisky scale is a validated scale designed to estimate the risk of medication non-adherence. The Scale of the total score ranges from 0 to 8. We only report a total score. For a reported scale,
  * Zero reflects worse medication adherence and
  * 8 reflects better medication adherence We didn't combine the subscales to compute a total score, but the total score does reflect the number of individual items that were endorsed.
Time Frame: 12 months minus baseline values
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Education and Lifestyle Coaching | Usual Care (UC) Control Arm
Number analyzed (Participants) | 49 | 48
score on a scale | 5.4 (2.3) | 4.6 (2.3)

ADVERSE EVENTS:
Time Frame: No adverse event data were collected over 12 month period of study intervention. There was no active monitoring for adverse events. However, upon completion of the study, our efforts to identify the reasons that led to study attrition, we found that a number of participants had passed away. None of the deaths were deemed to be a result of study participation.
Groups:
- Educational Intervention: Education and life style coaching includes:
  education about diabetes and kidney disease Coaching /counseling about lifestyle, nutrition and medication adherence
- Usual Care - Control: once randomize to the Usual Care control group, the participants are left alone and are suggested to contact their providers for health care. The group gets labs and other survey done at 6 and 12 months of the intervention.
Arm/Group | Educational Intervention | Usual Care - Control
All-Cause Mortality (participants affected / at risk) | 1/63 | 3/62
Serious Adverse Events (participants affected / at risk) | 1/63 | 3/62
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Educational Intervention (N=63) | Usual Care - Control (N=62)
Death (General disorders) | 1 | 3 — The causes of deaths were not known to us. So for that reason we listed it as General disorder
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Educational Intervention (N=0) | Usual Care - Control (N=0)
Other adverse event (General disorders) | 0 (0) | 0 (0) — We did not collect other adverse event

LIMITATIONS AND CAVEATS:
The study took place in one Indian reservation in rural New Mexico. The results might be different for people in other places. The team didn't look at which parts of the program might explain the changes they found.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No